CLINICAL TRIAL: NCT06642246
Title: Sleep Promotion Among Children Newly Diagnosed With Essential Hypertension
Brief Title: Sleep Promotion and Pediatric Hypertension
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 24-022262
Record Dates: First submitted 2024-10-04; First posted 2024-10-15 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Insufficient Sleep; Hypertension
Keywords: Insufficient Sleep; Hypertension
MeSH Terms: conditions — Sleep Deprivation; Hypertension | interventions — Methods

STUDY DESIGN:
Intervention Model Description: The study conditions are as follows: sleep goal, digital sleep guidance, loss-framed financial incentive, and personalized feedback. All participants need to self-monitor their sleep duration by wearing the sleep tracker to allow for daily capture of sleep duration and goal achievement status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Sleep goal, Sleep guidance messaging, Loss-framed incentive, Supportive feedback.
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Intervention — During a 7-week intervention phase, parent-child dyads will be provided a sleep duration goal paired with a loss-framed financial incentive (virtual account) starting with deductions each time the sleep goal is not met, will be sent sleep guidance text messages, and will receive weekly performance feedback text messages.

SUMMARY:
Determine the effectiveness and feasibility of a mobile health sleep extension approach in the pediatric nephrology setting, to increase sleep duration and reduce systolic and diastolic blood pressure.

DETAILED DESCRIPTION:
Insufficient sleep is associated with hypertension in children. Despite this knowledge, sleep promotion is not considered as a behavioral target during the initial treatment of pediatric essential hypertension. Investigators are developing a mobile platform to promote sleep in children that may have utility for treating pediatric essential hypertension.

The overall objective of this study is to determine the effectiveness and feasibility of a mobile health sleep extension approach in the pediatric nephrology setting, to increase sleep duration and reduce systolic and diastolic blood pressure.

This is a home-based, single-site study, of 13-to-18-year-olds (N=10, 5 parent-child dyads). Participants will have a recent diagnosis of essential hypertension, based on clinical ambulatory blood pressure monitoring, with initial treatment targeting lifestyle modification without pharmacological therapy. Participants must have cellular or internet access and spend less than or equal to 7.5 hours in bed per night. Children will be excluded if they have a known clinical sleep disorder.

The sleep promotion intervention will be delivered using REDCap. All participants will be provided with a sleep tracker to monitor their sleep patterns throughout the study. A two-week run-in phase will be used to capture baseline sleep patterns, and a home sleep polysomnography test will be completed to provide clinical sleep data. During a 7-week intervention phase, all participants will receive the same intervention condition. Participants will be provided a sleep duration goal paired with a loss-framed financial incentive (virtual account) starting with deductions each time the sleep goal is not met, will be sent sleep guidance text messages, and will receive weekly performance feedback text messages. Further, at the end of the intervention phase, participants will undergo a second Ambulatory Blood Pressure Monitoring (ABPM). The primary outcome is acceptance and feasibility of completing this study captured via self-reported feedback and documenting compliance with the study protocol. The secondary outcomes are changes in sleep duration from baseline, and changes in daytime and nocturnal systolic and diastolic blood pressure from baseline.

ELIGIBILITY:
Inclusion Criteria:

* Speak, read and write in English.
* Parental/guardian permission (informed consent) and child assent.
* Have a computer or a tablet computer with access to the Internet or own a smartphone with a data and text plan.
* Parent reported sleep duration on school nights less than or equal to 7.5 hours.
* Recently diagnosed with essential hypertension by Ambulatory Blood Pressure Monitoring (ABPM).
* If taking over the counter sleep aides, willing to stop them over the course of the study.

Exclusion Criteria:

* Any clinically diagnosed sleep disorder (e.g. sleep apnea) in the electronic health record and or regular use of prescribed sleep aide.
* Underlying chronic medical conditions, defined as a medical condition with a duration or expected duration longer than 3 months that involved taking regular medication, taking medications that could affect blood pressure (e.g., anti-hypertensive medications, glucocorticoids, or stimulants), and patients with underlying diagnoses known to be associated with elevated blood pressure (e.g., cardiac disease, kidney disease or diabetes).

Inclusion Criteria for Parents/Legal Guardians:

* Be the parent/guardian of an eligible child enrolled in the main study.
* Speak, read, and write in English.

Exclusion Criteria for Parents/Legal Guardians:

- Limited English proficiency

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Hypertension | From baseline to approximately week 11
  The number of participants who are still diagnosed with hypertension by ambulatory blood pressure monitoring (ABPM). This is defined as a mean systolic or diastolic blood pressure when either awake or asleep, greater than the 95th percentile.
Change in sleep tracker estimated weeknight sleep duration | From baseline to approximately week 11
  Change in sleep tracker estimated weeknight sleep duration will be measured from baseline (operationalized as the average hours per weeknight per week). There will be one week of baseline data and seven weeks of intervention data as well as two weeks of follow-up data.

SECONDARY OUTCOMES:
Change in sleep tracker estimated sleep duration | From baseline to approximately week 11
  Change in sleep tracker estimated sleep duration will be measured from baseline (operationalized as the average hours per night per week). There will be one week of baseline data and seven weeks of intervention data as well as two weeks of follow-up data.
Changes in sleep disturbance score measured by the Patient-Reported Outcome Measurement System (PROMIS) tool | From baseline to approximately week 11
  Measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) item bank for pediatric sleep. This validated survey generates a composite sleep disturbance T-score based on items related to sleep onset, sleep continuity and sleep quality in the past week. Higher T-scores indicates poorer sleep quality.
Change in daytime systolic/diastolic blood pressures as measured by Ambulatory Blood Pressure Monitoring (ABPM) | From baseline to approximately week 11
  Changes in daytime systolic and diastolic blood pressure from baseline. Measured variables include daytime systolic/diastolic mean BP, BP index (calculated by dividing the average BP of the participant by the sex and height specific 95th percentiles for systolic and diastolic BP].
Change in night time systolic/diastolic blood pressures as measured by ABPM | From baseline to approximately week 11
  Changes in nocturnal systolic and diastolic blood pressure from baseline. Measured variables include nighttime systolic/diastolic mean BP, percent nocturnal dipping, BP index (calculated by dividing the average BP of the participant by the sex and height specific 95th percentiles for systolic and diastolic BP].

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Mitchell, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sadeh A, Gruber R, Raviv A. The effects of sleep restriction and extension on school-age children: what a difference an hour makes. Child Dev. 2003 Mar-Apr;74(2):444-55. doi: 10.1111/1467-8624.7402008. PMID 12705565
- [Background] Mindell JA, Sedmak R, Boyle JT, Butler R, Williamson AA. Sleep Well!: A Pilot Study of an Education Campaign to Improve Sleep of Socioeconomically Disadvantaged Children. J Clin Sleep Med. 2016 Dec 15;12(12):1593-1599. doi: 10.5664/jcsm.6338. PMID 27655459
- [Background] Meltzer LJ, Williamson AA, Mindell JA. Pediatric sleep health: It matters, and so does how we define it. Sleep Med Rev. 2021 Jun;57:101425. doi: 10.1016/j.smrv.2021.101425. Epub 2021 Jan 19. PMID 33601324
- [Background] Allen SL, Howlett MD, Coulombe JA, Corkum PV. ABCs of SLEEPING: A review of the evidence behind pediatric sleep practice recommendations. Sleep Med Rev. 2016 Oct;29:1-14. doi: 10.1016/j.smrv.2015.08.006. Epub 2015 Sep 1. PMID 26551999
- [Background] Mitchell JA, Morales KH, Williamson AA, Jawahar A, Juste L, Vajravelu ME, Zemel BS, Dinges DF, Fiks AG. Promoting Sleep Duration in the Pediatric Setting Using a Mobile Health Platform: A Randomized Optimization Trial. medRxiv [Preprint]. 2023 Jan 5:2023.01.04.23284151. doi: 10.1101/2023.01.04.23284151. PMID 36711634
- [Background] Mitchell JA, Morales KH, Williamson AA, Huffnagle N, Eck C, Jawahar A, Juste L, Fiks AG, Zemel BS, Dinges DF. Engineering a mobile platform to promote sleep in the pediatric primary care setting. Sleep Adv. 2021 Apr 15;2(1):zpab006. doi: 10.1093/sleepadvances/zpab006. eCollection 2021. PMID 33981997
- [Background] Tversky A, Kahneman D. The framing of decisions and the psychology of choice. Science. 1981 Jan 30;211(4481):453-8. doi: 10.1126/science.7455683.
- [Background] Chokshi NP, Adusumalli S, Small DS, Morris A, Feingold J, Ha YP, Lynch MD, Rareshide CAL, Hilbert V, Patel MS. Loss-Framed Financial Incentives and Personalized Goal-Setting to Increase Physical Activity Among Ischemic Heart Disease Patients Using Wearable Devices: The ACTIVE REWARD Randomized Trial. J Am Heart Assoc. 2018 Jun 13;7(12):e009173. doi: 10.1161/JAHA.118.009173. PMID 29899015
- [Background] Patel MS, Asch DA, Rosin R, Small DS, Bellamy SL, Heuer J, Sproat S, Hyson C, Haff N, Lee SM, Wesby L, Hoffer K, Shuttleworth D, Taylor DH, Hilbert V, Zhu J, Yang L, Wang X, Volpp KG. Framing Financial Incentives to Increase Physical Activity Among Overweight and Obese Adults: A Randomized, Controlled Trial. Ann Intern Med. 2016 Mar 15;164(6):385-94. doi: 10.7326/M15-1635. Epub 2016 Feb 16. PMID 26881417
- [Background] Long JA, Jahnle EC, Richardson DM, Loewenstein G, Volpp KG. Peer mentoring and financial incentives to improve glucose control in African American veterans: a randomized trial. Ann Intern Med. 2012 Mar 20;156(6):416-24. doi: 10.7326/0003-4819-156-6-201203200-00004. PMID 22431674
- [Background] Sen AP, Sewell TB, Riley EB, Stearman B, Bellamy SL, Hu MF, Tao Y, Zhu J, Park JD, Loewenstein G, Asch DA, Volpp KG. Financial incentives for home-based health monitoring: a randomized controlled trial. J Gen Intern Med. 2014 May;29(5):770-7. doi: 10.1007/s11606-014-2778-0. Epub 2014 Feb 13. PMID 24522623
- [Background] Volpp KG, John LK, Troxel AB, Norton L, Fassbender J, Loewenstein G. Financial incentive-based approaches for weight loss: a randomized trial. JAMA. 2008 Dec 10;300(22):2631-7. doi: 10.1001/jama.2008.804. PMID 19066383
- [Background] Kuna ST, Shuttleworth D, Chi L, Schutte-Rodin S, Friedman E, Guo H, Dhand S, Yang L, Zhu J, Bellamy SL, Volpp KG, Asch DA. Web-Based Access to Positive Airway Pressure Usage with or without an Initial Financial Incentive Improves Treatment Use in Patients with Obstructive Sleep Apnea. Sleep. 2015 Aug 1;38(8):1229-36. doi: 10.5665/sleep.4898. PMID 25581921
- [Background] Wong CA, Miller VA, Murphy K, Small D, Ford CA, Willi SM, Feingold J, Morris A, Ha YP, Zhu J, Wang W, Patel MS. Effect of Financial Incentives on Glucose Monitoring Adherence and Glycemic Control Among Adolescents and Young Adults With Type 1 Diabetes: A Randomized Clinical Trial. JAMA Pediatr. 2017 Dec 1;171(12):1176-1183. doi: 10.1001/jamapediatrics.2017.3233. PMID 29059263
- [Background] Asch DA, Troxel AB, Stewart WF, Sequist TD, Jones JB, Hirsch AG, Hoffer K, Zhu J, Wang W, Hodlofski A, Frasch AB, Weiner MG, Finnerty DD, Rosenthal MB, Gangemi K, Volpp KG. Effect of Financial Incentives to Physicians, Patients, or Both on Lipid Levels: A Randomized Clinical Trial. JAMA. 2015 Nov 10;314(18):1926-35. doi: 10.1001/jama.2015.14850. PMID 26547464
- [Background] Mullins EN, Miller AL, Cherian SS, Lumeng JC, Wright KP Jr, Kurth S, Lebourgeois MK. Acute sleep restriction increases dietary intake in preschool-age children. J Sleep Res. 2017 Feb;26(1):48-54. doi: 10.1111/jsr.12450. Epub 2016 Sep 19. PMID 27641365
- [Background] Simon SL, Field J, Miller LE, DiFrancesco M, Beebe DW. Sweet/dessert foods are more appealing to adolescents after sleep restriction. PLoS One. 2015 Feb 23;10(2):e0115434. doi: 10.1371/journal.pone.0115434. eCollection 2015. PMID 25706861
- [Background] Beebe DW, Fallone G, Godiwala N, Flanigan M, Martin D, Schaffner L, Amin R. Feasibility and behavioral effects of an at-home multi-night sleep restriction protocol for adolescents. J Child Psychol Psychiatry. 2008 Sep;49(9):915-23. doi: 10.1111/j.1469-7610.2008.01885.x. Epub 2008 Jun 28. PMID 18564072
- [Background] Van Dyk TR, Zhang N, Catlin PA, Cornist K, McAlister S, Whitacre C, Beebe DW. Feasibility and Emotional Impact of Experimentally Extending Sleep in Short-Sleeping Adolescents. Sleep. 2017 Sep 1;40(9). doi: 10.1093/sleep/zsx123. PMID 28934531
- [Background] Van Dyk TR, Krietsch KN, Saelens BE, Whitacre C, McAlister S, Beebe DW. Inducing more sleep on school nights reduces sedentary behavior without affecting physical activity in short-sleeping adolescents. Sleep Med. 2018 Jul;47:7-10. doi: 10.1016/j.sleep.2018.03.007. Epub 2018 Mar 29. PMID 29880148
- [Background] Hart CN, Carskadon MA, Considine RV, Fava JL, Lawton J, Raynor HA, Jelalian E, Owens J, Wing R. Changes in children's sleep duration on food intake, weight, and leptin. Pediatrics. 2013 Dec;132(6):e1473-80. doi: 10.1542/peds.2013-1274. Epub 2013 Nov 4. PMID 24190680
- [Background] Beebe DW, Simon S, Summer S, Hemmer S, Strotman D, Dolan LM. Dietary intake following experimentally restricted sleep in adolescents. Sleep. 2013 Jun 1;36(6):827-34. doi: 10.5665/sleep.2704. PMID 23729925
- [Background] Gruber R, Cassoff J, Frenette S, Wiebe S, Carrier J. Impact of sleep extension and restriction on children's emotional lability and impulsivity. Pediatrics. 2012 Nov;130(5):e1155-61. doi: 10.1542/peds.2012-0564. Epub 2012 Oct 15. PMID 23071214
- [Background] Fobian AD, Elliott L, Louie T. A Systematic Review of Sleep, Hypertension, and Cardiovascular Risk in Children and Adolescents. Curr Hypertens Rep. 2018 May 1;20(5):42. doi: 10.1007/s11906-018-0841-7. PMID 29717377
- [Background] Williams JA, Zimmerman FJ, Bell JF. Norms and trends of sleep time among US children and adolescents. JAMA Pediatr. 2013 Jan;167(1):55-60. doi: 10.1001/jamapediatrics.2013.423. PMID 23403646
- [Background] Matricciani LA, Olds TS, Blunden S, Rigney G, Williams MT. Never enough sleep: a brief history of sleep recommendations for children. Pediatrics. 2012 Mar;129(3):548-56. doi: 10.1542/peds.2011-2039. Epub 2012 Feb 13. PMID 22331340
- [Background] Paruthi S, Brooks LJ, D'Ambrosio C, Hall WA, Kotagal S, Lloyd RM, Malow BA, Maski K, Nichols C, Quan SF, Rosen CL, Troester MM, Wise MS. Consensus Statement of the American Academy of Sleep Medicine on the Recommended Amount of Sleep for Healthy Children: Methodology and Discussion. J Clin Sleep Med. 2016 Nov 15;12(11):1549-1561. doi: 10.5664/jcsm.6288. PMID 27707447